CLINICAL TRIAL: NCT04986189
Title: Lung Screening for Hodgkin Lymphoma Survivors: a Feasibility Study
Brief Title: Lung Screening in People Cured of Hodgkin Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CFTSp204
Record Dates: First submitted 2021-05-26; First posted 2021-08-02 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Hodgkin Lymphoma; Lung Cancer
Keywords: screening; low dose CT scan
MeSH Terms: conditions — Hodgkin Disease; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Invitation to have a low dose CT thorax (Other): All participants are invited to undergo a low dose CT thorax
  Interventions: Diagnostic Test: Low dose CT thorax

INTERVENTIONS:
Diagnostic Test: Low dose CT thorax — A low dose CT scan of the thorax to screen for lung cancer

SUMMARY:
A single site non-commercial study in which people treated for Hodgkin lymphoma survivors will be invited to have a single low dose CT of thorax for lung cancer screening

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80
* 5 year or more survivor of HL
* Any of: a) treated with radiotherapy for HL with radiation dose to the lung b) an alkylating agent containing chemotherapy regimen known to increase lung cancer risk
* Living within approximately 40 miles of The Christie Hospital

Exclusion Criteria:

* Previous diagnoses of malignant neoplasm of trachea, bronchus, lung, thymus or pleura
* A current diagnosis of metastatic cancer
* Residents in nursing homes or housebound
* Had a CT scan of the thorax within the last 12 months
* Pregnant women
* Unable to provide consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Primary outcome: the lung cancer screening uptake rate among eligible individuals invited to the study | Measured 6 months after recruitment begins when all interested participants have undergone a full eligibility check and those eligible have undergone their baseline low dose CT scan
  Feasibility outcome

SECONDARY OUTCOMES:
Decisional conflict scores in those who receive the decision aid measured using the validated Decisional Conflict Scale (score 0-100 with higher score representing higher levels of decisional conflict) | 14 months
Preparedness for decision making in those who receive the decision aid using the validated Preparedness for Decision Making Scale (score 0-100 with higher score representing higher perceived levels of preparedness for decision making) | 4 months
Lung cancer screening knowledge pre and post receipt of the decision aid measured using a novel scale (score 0-16 with higher score representing high levels of knowledge about lung cancer screening) | 4 months
The proportion who have made an informed decision as measured by the Multidimensional Measure of Informed Choice | 6 and 12 months following CT scan
Anxiety levels pre and post screening measured using the State Trait Anxiety Inventory -6 validated scale (score 6-24 with higher score representing higher levels of anxiety) | 2 months post CT scan
Cancer worry severity levels pre and post screening measured using measured using 4-item Brief Worry Scale (score 4-20 with higher score representing higher cancer worry severity levels) | 12 months
Cancer worry frequency measured using intrusive thoughts subscale from Revised impact of events scale (score 6-30 with higher score representing more frequent cancer worry) | 12 months
Health related quality of life pre-screening then 6 and 12 months post screening measured using the validated SF-12 (short-form-12) scale (Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning) | 12 months
The rates of smoking cessation 6 and 12 months following screening | 12 months
The acceptability of undergoing screening measured using non-validated scale (Score 7-70 with higher score representing higher perceived acceptability of lung cancer screening) | 2 months
Rates of normal, indeterminate and positive screening scans, reported according to definitions in the British Thoracic Society Pulmonary Nodule Management Guidelines | 12 months
The type and prevalence of incidental findings on screening scans | 12 months
The barriers and facilitators to undergoing lung cancer screening measured qualitatively and categorised according to the Theoretical Domains Framework | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

REFERENCES:
- [Derived] Broadbent R, Crosbie P, Armitage CJ, Taylor B, Tenant S, Mercer J, Radford J, Linton K. Pilot study of lung cancer screening for survivors of Hodgkin lymphoma. Haematologica. 2024 Oct 1;109(10):3305-3313. doi: 10.3324/haematol.2023.283287. PMID 37981893